CLINICAL TRIAL: NCT03458507
Title: Impact of the Type of Interface in Neuromuscular Patients Treated With Nocturnal Noninvasive Ventilation: a Randomized Crossover Trial
Brief Title: Impact of the Type of Interface in Neuromuscular Patients Treated With Nocturnal Noninvasive Ventilation
Acronym: InterfaceNMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); Hôpital Raymond Poincaré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC17.346
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Neuromuscular Diseases; Alveolar Hypoventilation
Keywords: Neuromuscular diseases; Non-invasive ventilation; Nasal mask; Oronasal mask; Alveolar hypoventilation; leaks; Sleep disorder breathing; Side effects
MeSH Terms: conditions — Neuromuscular Diseases; Hypoventilation

STUDY DESIGN:
Intervention Model Description: The patients will be randomized for two periods of one week to use NIV either with nasal or oronasal mask. The randomization will be stratified according to the type of interface previously used at home by the patient (nasal and oronasal). Such stratification will allow a balance between the number of patients that will begin with their usual interface versus with an alternative interface. In these patients, NIV withdrawal is not acceptable in terms of patient's security and ethics. Therefore, it is not possible to include a wash out period between both arms. The potential carry-over effect will be taken into account in the statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual interface (Active Comparator): Patients which begin with their usual interface for one week, home polygraphy and side effect assessment at the end of the first week.
  Switch for alternative interface, seven days familiarisation, second polygraphy and side effect assessment at the end of the second week.
  Interventions: Device: Switch of nocturnal NIV interface
- Alternative interface (Active Comparator): Patients which begin with the alternative interface for one week, home polygraphy and side effect assessment at the end of the first week.
  Switch for usual interface, seven days with usual device, second polygraphy and side effect assessment at the end of the second week.
  Interventions: Device: Switch of nocturnal NIV interface

INTERVENTIONS:
Device: Switch of nocturnal NIV interface — 1. test the alternative interfaces (either a nasal mask for the patient used to oronasal mask or inversely an oronasal mask if the usual mask is nasal) during a one-hour diurnal NIV session. SpO2 (polygraphy), PtcCO2 will be monitored continuously during this diurnal session. Patients will use their usual NIV device prescribed at home. NIV settings will be adapted if needed.
  2. Interface switch
  3. unattended nocturnal polygraphy under NIV (cf details below) will be performed at home with SomnoHolter® (Nomics, Liege, Belgium), synchronized with transcutaneous partial pressure in CO2 (PtcCO2) monitoring by SenTec V-Sign™ System.
  The PtcCO2 device will be calibrated before and at the end of each night to allow drift correction.

SUMMARY:
Nocturnal Non Invasive Ventilation (NIV) is the reference treatment for chronic alveolar hypoventilation in patients with neuro-muscular diseases. NIV can be provided by using different types of interfaces: Nasal masks are the most frequent type of interface used at home but oronasal masks are used by at least 25% of neuro-muscular patients mainly because of persistent unintentional mouth leaks. However, oronasal mask may cause persistent upper airway obstructive respiratory events because of the mechanical constraint on the chin induced by the traction of the straps that may push the mandible posteriorly during sleep.

No randomized study has specifically addressed the question of the impact of type of interface in patients with neuromuscular diseases treated by nocturnal NIV.

The investigators hypothesize that:

1. the application of oronasal mask may jeopardize the pharyngeal patency in patients already proned to upper airway obstruction;
2. the use of a nasal mask may improve upper airway stability and NIV efficacy while reducing side effects.

Authors objective will be to compare the impact of nasal mask versus oronasal mask on NIV efficacy and side-effects. Eligible patients are those with nocturnal NIV and neuromuscular disease.

After a scheduled hospital visit, patients willing to participate will undergo in random order 2 unattended nocturnal polygraphies under NIV at home: one polygraphy with nasal mask; one with an oronasal mask. Each polygraphy ans side effects assessment will be performed after one week of familiarization with each mask.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Affected by slowly progressive neuro-muscular diseases (Becker muscular dystrophy, facio-scapulo-humeral dystrophy, limb-girdle dystrophy, myotonic dystrophy…) or relatively rapid progression (Duchenne muscular dystrophy).
* Treated with nocturnal non-invasive ventilation (<15 hours/day)
* In stable state (no cardiorespiratory or ear-nose-throat event for at least 1 month before inclusion)

Exclusion Criteria:

* Rapidly progressive neuro-muscular diseases (such as ALS)
* Severe nasal obstruction, maxillofacial deformities or previous upper airway surgery preventing the usage of one type of mask (nasal or oronasal), or, at the discretion of investigator, any other contraindication for using the other type of mask
* NIV Daily use >15h/day
* Unwillingness or inability to provide consent to participation
* Curatorship
* Subject in exclusion period of another study
* Vulnerable person or legally protected adult.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Mean nocturnal oxygen saturation (SpO2) | After one week with each type of mask
  Mean nocturnal SpO2, measured by oximetry.

SECONDARY OUTCOMES:
% sleep recording with SpO2<90% | After one week with each type of mask
  Percentage of sleep recording spent with SpO2<90% between oronasal mask versus nasal mask
Oxygen Desaturation Index | After one week with each type of mask
  Oxygen desaturation index between oronasal mask versus nasal mask
Mean nocturnal PtcCO2 | After one week with each type of mask
  Mean nocturnal transcutaneous partial pressure in CO2 (PtcCO2) evaluated by capnography between oronasal mask versus nasal mask
Mean mouth opening during sleep | After one week with each type of mask
  Mean mouth opening during sleep between oronasal mask versus nasal mask
Non-intentional leaks | After one week with each type of mask
  Non-intentional leaks recorded by the NIV-device
Side-effects of Continuous Positive Airway Pressure (CPAP) | After one week with each type of mask
  Side-effects reported by patients using a modified version of "Side Effect of CPAP inventory" (SECI) questionnaire.
  A French translation will be done by two bilingual investigators (one medical doctor, one linguist).
  This questionnaire consists of a list of 15 commonly reported side effects under CPAP.
  For each side effect, the patient is asked to rate the frequency (0-5), magnitude (0-5) and perceived impact on adherence (0-5) on a five-point Likert-type scale.
  Total score range : 0 to 225, with the higher score associated with the worst tolerance.
  Range for each of the fifteen side effects: 0 to 15, higher values always represent a worse outcome (all subscales results are summed to compute the total score)

CONTACTS AND LOCATIONS:
Locations (1):
- Grenoble-Alpes University hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borel JC, Tamisier R, Dias-Domingos S, Sapene M, Martin F, Stach B, Grillet Y, Muir JF, Levy P, Series F, Pepin JL; Scientific Council of The Sleep Registry of the French Federation of Pneumology (OSFP). Type of mask may impact on continuous positive airway pressure adherence in apneic patients. PLoS One. 2013 May 15;8(5):e64382. doi: 10.1371/journal.pone.0064382. Print 2013. PMID 23691209
- [Background] Bakker JP, Neill AM, Campbell AJ. Nasal versus oronasal continuous positive airway pressure masks for obstructive sleep apnea: a pilot investigation of pressure requirement, residual disease, and leak. Sleep Breath. 2012 Sep;16(3):709-16. doi: 10.1007/s11325-011-0564-3. Epub 2011 Jul 29. PMID 21800222
- [Background] Borel JC, Gakwaya S, Masse JF, Melo-Silva CA, Series F. Impact of CPAP interface and mandibular advancement device on upper airway mechanical properties assessed with phrenic nerve stimulation in sleep apnea patients. Respir Physiol Neurobiol. 2012 Aug 15;183(2):170-6. doi: 10.1016/j.resp.2012.06.018. Epub 2012 Jul 3. PMID 22772315
- [Background] Willson GN, Piper AJ, Norman M, Chaseling WG, Milross MA, Collins ER, Grunstein RR. Nasal versus full face mask for noninvasive ventilation in chronic respiratory failure. Eur Respir J. 2004 Apr;23(4):605-9. doi: 10.1183/09031936.04.00051604. PMID 15083762
- [Background] Fleck RJ Jr, Mahmoud M, McConnell K, Shott SR, Gutmark E, Amin RS. An adverse effect of positive airway pressure on the upper airway documented with magnetic resonance imaging. JAMA Otolaryngol Head Neck Surg. 2013 Jun;139(6):636-8. doi: 10.1001/jamaoto.2013.3279. PMID 23787424
- [Background] Vrijsen B, Buyse B, Belge C, Testelmans D. Upper airway obstruction during noninvasive ventilation induced by the use of an oronasal mask. J Clin Sleep Med. 2014 Sep 15;10(9):1033-5. doi: 10.5664/jcsm.4046. PMID 25142771
- [Derived] Leotard A, Delorme M, Hartley S, Khouri C, Lebret M, Lofaso F, Pepin JL, Borel JC. Non-invasive ventilation in neuromuscular diseases: should we use higher levels of ventilatory support? Sleep Breath. 2023 May;27(2):673-677. doi: 10.1007/s11325-022-02658-3. Epub 2022 Jun 20. PMID 35725863
- [Derived] Leotard A, Lebret M, Daabek N, Prigent H, Destors M, Saint-Raymond C, Sagniez A, Leroux K, Tamisier R, Lofaso F, Pepin JL, Borel JC. Impact of Interface Type on Noninvasive Ventilation Efficacy in Patients With Neuromuscular Disease: A Randomized Cross-Over Trial. Arch Bronconeumol (Engl Ed). 2021 Apr;57(4):273-280. doi: 10.1016/j.arbres.2020.05.024. Epub 2020 Jun 23. English, Spanish. PMID 32586702